CLINICAL TRIAL: NCT01399437
Title: Default Network Dysfunction Underlying Visuospatial Attention Deficits in Schizophrenia
Brief Title: Brain Functions Underlying Visuospatial Attention Deficits in Schizophrenia
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911470; 11-DA-N470
Record Dates: First submitted 2011-07-20; First posted 2011-07-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2014-12-24

CONDITIONS: Schizophrenia
Keywords: Default Network; Schizophrenia; fMRI; Spatial Attention; Sentinel Function
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- A special brain circuit is important for helping us keeping an eye open for things that are going on around us, even when we are not directly paying attention to them. This circuit seems to work differently in people with schizophrenia than in other people, which may explain specific deficits with broad monitoring observed in people with schizophrenia. Researchers want to compare brain function in people with schizophrenia and healthy volunteers to find out more about how these brain circuits work and affect attention.

Objectives:

- To study how the brain performs broad visual monitoring in people with schizophrenia.

Eligibility:

* Individuals between 18 to 55 years of age who have been diagnosed with schizophrenia.
* Healthy volunteers between 18 and 55.

Design:

* Participants will be screened with physical and psychological exams. They will have a medical history. Tests for drug and alcohol use will also be done.
* Participants will have two study visits. The first is a training visit and the second is a scanning visit.
* At the training visit, participants will practice computer-based tests of focus, memory, and concentration. They will also answer questions about mood, psychiatric symptoms, and smoking habits.
* At the scanning visit, participants will perform the computer-based tasks that they practiced at the training visit. They will have magnetic resonance imaging while they perform these tasks.

DETAILED DESCRIPTION:
Objective: To test a neural circuit explanation for a visuospatial attention abnormality seen in schizophrenia. Specifically, the aim is to test whether broad monitoring deficits may be based on a disruption of the so-called sentinel function of the default network. Because the default network is modulated by nicotinic compounds, such finding would implicate a possible remediation strategy.<TAB>

Study population: 24 people with schizophrenia, 24 matched healthy control subjects.

Design: A group comparison of attention task performance and associated brain activity as measured by functional Magnetic Resonance Imaging.

Outcome measures: Measures of attention task performance (reaction time, accuracy), BOLD signal within regions of the default network, degree of temporal association of BOLD signal with trial-by-trial reaction time.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants:

1. Age 18 through 55.
2. Normal or corrected to normal visual acuity (at least 20/80)

   Participants with menat illness:
3. DSM-IV diagnosis of schizophrenia or schizoaffective disorder
4. Ability to give written informed consent
5. Four week of stable pharmacological treatment (same psychiatric medication at same dose or no medication)

EXCLUSION CRITERIA:

All participants:

1. Presence of ferromagnetic metal objects in the body, implanted electronic devices or any other counter -indication for MRI.
2. Claustrophobia
3. Left handed or ambidextrous
4. History of myocardial infarction or heart failur, which may cause asymptomatic brain lesions
5. Uncontrolled high blood pressure (resting systolic greater than 150 or diastolic greater than 90 mm Hg)
6. Neurological conditions likely to impair cognitive function such as stroke, seizures, dementia or organic brian syndrome
7. Any condition likely to impair cognitive function such as mental retardation or severe pharmacological sedation
8. Current use of vasodilating beta-blockers (carvedilol, labetalol or nebivolol)
9. Alcohol or substance abuse or dependence other than nicotine within the last 6 months
10. Pregnancy, verified by urin pregnancy test for females during screening and on the day of the scan.

    Healthy Controls:
11. Current psychiatric Axis I disorder or Axis II schizophrenia spectrum disorder, verified by Structured Clinical Interview for DSM-IV (SCID)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-07-03; Study Completion 2014-12-24

PRIMARY OUTCOMES:
Behavioral performance measures on the cognitive tasks (e.g. reaction time, accuracy)
Bold signal, specifically activation of the default network of resting brain function and its association with task performance.

SECONDARY OUTCOMES:
Secondary outcome measures include ratings and scores on questionnaires and characterization tools.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- Maryland Psychiatric Research Center (MPRC) 55 Wade Avenue, Catonsville, Maryland, United States

REFERENCES:
- [Background] Binder JR, Frost JA, Hammeke TA, Bellgowan PS, Rao SM, Cox RW. Conceptual processing during the conscious resting state. A functional MRI study. J Cogn Neurosci. 1999 Jan;11(1):80-95. doi: 10.1162/089892999563265. PMID 9950716
- [Background] Buckner RL, Andrews-Hanna JR, Schacter DL. The brain's default network: anatomy, function, and relevance to disease. Ann N Y Acad Sci. 2008 Mar;1124:1-38. doi: 10.1196/annals.1440.011. PMID 18400922
- [Background] Bustillo JR, Thaker G, Buchanan RW, Moran M, Kirkpatrick B, Carpenter WT Jr. Visual information-processing impairments in deficit and nondeficit schizophrenia. Am J Psychiatry. 1997 May;154(5):647-54. doi: 10.1176/ajp.154.5.647. PMID 9137120